CLINICAL TRIAL: NCT03216941
Title: Prospective Randomised Double Blind Trial of Ketiapine and Olanzapine Comparative Efficacy for Fast Sedation of Severely Agitated Patients in Emergency Psychiatric Ward
Brief Title: Randomised Trial Ketiapine Olanzapine Fast Sedation Agitated Patients Emergency Ward
Acronym: IM-OK-FAST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad Nacional de Rosario (Other)
Responsible Party: Principal Investigator, daniel serrani, Dr, Universidad Nacional de Rosario
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: msm1
Record Dates: First submitted 2017-07-10; First posted 2017-07-13 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Psychomotor Agitation; Psychiatric Disorder; Emergency Psychiatric; Tranquilizers
Keywords: Psychomotor agitation; Tranquilizing agents
MeSH Terms: conditions — Psychomotor Agitation; Mental Disorders | interventions — Ketamine; Olanzapine

STUDY DESIGN:
Intervention Model Description: double-blind controlled trial to compare the effectiveness of intramuscular olanzapine and ketamine as first medication(s) used to treat patients with agitation caused by psychosis.
Who Masked: Care Provider
Masking Description: care provider were masked with regard to the patient's treatment assignment, and patients were instructed not to reveal their current treatment to the investigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketamine (Active Comparator): assessment of agitation status with Ramsay Sedation Scale administration of ketamine 10 mg / ml IM one dose supervision of vital signs registration of time of ketamine administration registration of time when expected outcome is obtained follow up of vital signs supervision until obsevation period expires (12 hours after admission to emergency board) registration of adverse effects registration if other interventions were applied (aside of ketamine administration) withdrawal of patient from the study if other medication was needed (aside of ketamine)
  Interventions: Drug: Ketamine
- olanzapine (Active Comparator): assessment of agitation status with Ramsay Sedation Scale administration of olanzapine 10 mg / ml IM one dose supervision of vital signs registration of time of olanzapine administration registration of time when expected outcome is obtained follow up of vital signs supervision until obsevation period expires (12 hours after admission to emergency board) registration of adverse effects registration if other interventions were applied (aside of olanzapine administration) withdrawal of patient from the study if other medication was needed (aside of olanzapine)
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — study medications were packaged in identical color-coded boxes. first dosage included either 10 mg of olanzapine, or 10 mg of ketamine Dosages were chosen based on previous studies After the initial dose, no additional dosis were allowed if supplemental medication eas needed according to clinician judgment the subject will be immediately removed from the study.
  All subjects will be assessed 1 hour, 2 hours, 4 hours, 6 hours and 12 hours after t he first administration of the medication.
  Other Names: olanzapine

SUMMARY:
comparison of intramuscular olanzapine and ketamine efficacy as first medication for fast sedation of patients with agitation and aggressive behavior. Five hundred patients with agitation caused by psychiatric disorder were randomly assigned under double-blind conditions to receive olanzapine or ketiapine. The Overt Agitation Severity Scale, Overt Aggression Scale and Ramsay Sedation Scale will be applied within 12 hours after the first dosage.

DETAILED DESCRIPTION:
double-blind controlled trial to compare effectiveness of intramuscular olanzapine and ketamine as first medication to fast sedation of patients with agitation caused by psychiatric conditions. Randomization will be performed by permuted blocks allocation in which ketiamine or olanzapine standard treatment will be assigned to blocks of five patients and distributed in this order: olanzapine and ketiamine. This assignment will be repeated until the total number of subjects (500) be reached.

agitation status will be operationalized using Overt Agitation Severity Scale Total Score (OASS) equal or greater than 20 and Overt Aggressive Scale (OAS) with four or more positive items. Full physical and neurological examination will be completed as soon as possible, whenever patient is considered eligible for the study. Written Informed consent should be provided before and after participating in this study, and should be reviewed and approved by the institutional review board. Written consent obtained before admission to the emergency ward by legal guardian and after 12 hours by the patient (whenever he or she is is able to understand the information) or by the guardian. This study will comply with principles of the Declaration of Helsinki and Good Clinical Practice and approved by the Institutional Review Board (IRB) of Hospital Larcade of San Miguel County (Province of Buenos AIres (Project msm001) inter-rater reproducibility will be evaluated by two raters which will repeatedly apply OASS, OAS and RSS to patients admitted to the emergency room before the study until the intraclass correlation coefficient (ICC) reach a score of 0.80 or greater medications will be packaged in identical color-coded boxes and dosage of of olanzapine and ketiamine will be determined according to standard protocols and previous studies.

If a subject needs another intervention will be removed from the study. subjects will be assessed from 1 to 12 hours after administration of selected medication.

psychiatrists will be masked to patient's treatment assignment, and patients will be instructed not to reveal current treatment to investigators.

clinical safety of treatment will be assessed by notification and with an close-ended inquiry into adverse events together with full physical examination and vital signs measurements. Statistical analyses mean and standard deviation (SD) and comparisons of baseline demographic and clinical characteristics with one-way analysis of variance (ANOVA), chi-square test for categorical variables and mixed-effect analyses of covariance (ANCOVAs) with medication (olanzapine, ketiamine) as between-groups factor and time (1 hour, 2 hours, 4 hours, 6 hours and 12 hours) as a within-group factor. OASS at time zero, OAS at time zero, and presence of excessive sedation will be fixe covariates, and symptom ratings (OASS, OAS and RSS) will be time-varying covariates.

differences between groups at each time point and variance with post-hoc Duncan's tests will be calculated to compare mean OASS, OAS and RSS scores between groups.

ELIGIBILITY:
Inclusion Criteria:

* signs of agitation,
* age between 18 and 64 years,
* bipolar (maniac or mixed episode)
* psychotic disorder diagnosis
* disorders due to drug abuse,
* organic disorder,
* anxiety or personality disorder
* Overt Agitation Severity Scale Total Score (OASS) equal or greater than 20
* Overt Aggressive Scale (OAS) with four or more positive items.

Exclusion Criteria:

* failure to agree to participate in the study,
* incapability of completing all steps
* unstable clinical disease -
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2016-01-31 (Actual)

PRIMARY OUTCOMES:
sedation status | 1 to 12 hours
  subjects will be assessed 1 hour, 2 hours, 4 hours, 6 hours and 12 hours after administration of the medication with Ramsay Sedation Scale score (RSS).

SECONDARY OUTCOMES:
adverse effects | 1 to 24 hours
  extrapirarmidal effects with Angus Scale for extrapiramidal movements excessive sedation with Ramsay Sedation Scale score paradoxical agitation with Ramsay Sedation Scale Score

CONTACTS AND LOCATIONS:
Locations (1):
- hospital Larcade, San Miguel, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided
make accesible patients data on SPSS file formats with not personal ID data